CLINICAL TRIAL: NCT00940966
Title: A Pilot Study to Determine the Efficacy of a Low Carbohydrate Diet in Treatment of Adolescents With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Steven sondike MD, WVU department of pediatrics
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-02-1776
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Elevated Triglycerides; Systolic Hypertension; Insulin Resistance; Abdominal Obesity
Keywords: ADA diet; low carbohydrate diet; Metabolic syndrome
MeSH Terms: conditions — Hypertriglyceridemia; Isolated Systolic Hypertension; Insulin Resistance; Obesity, Abdominal; Metabolic Syndrome | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- energy restricted very-low carbohydrate (Experimental): non-energy restricted ketogenic diet .
  Interventions: Dietary Supplement: energy restricted very-low carbohydrate diet
- ADA diet (Active Comparator): standard ADA diet
  Interventions: Dietary Supplement: standard ADA diet; Dietary Supplement: energy restricted very-low carbohydrate diet
- low glycemic index (Active Comparator): restricted ketogenic diet
  Interventions: Dietary Supplement: low glycemic diet

INTERVENTIONS:
Dietary Supplement: standard ADA diet — standard ADA diet
  Arms: ADA diet
Dietary Supplement: energy restricted very-low carbohydrate diet — energy restricted very-low carbohydrate diet
  Arms: ADA diet; energy restricted very-low carbohydrate
Dietary Supplement: low glycemic diet — restricted ketogenic diet
  Other Names: ketogenic diet.
  Arms: low glycemic index

SUMMARY:
The purpose of this study is to determine the effectiveness of two different non-energy restricted controlled carbohydrate programs with the American Diabetes Associations' diet on glycosylated hemoglobin and other diabetes risk factors in obese adolescents with metabolic syndrome, a constellation of symptoms associated with the development of type 2 diabetes and cardiovascular disease.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of two different non-energy restricted controlled carbohydrate programs with the American Diabetes Associations' diet on glycosylated hemoglobin and other diabetes risk factors in obese adolescents with metabolic syndrome, a constellation of symptoms associated with the development of type 2 diabetes and cardiovascular disease.

We plan to address the following issues:

1. To test the hypothesis that a controlled carbohydrate nutrition plan will be superior to the standard ADA diet in controlling blood sugar (as measured by glycosylated hemoglobin [HbA1C]), decreasing cardiovascular risk factors (Serum Lipid Levels, Blood Pressure) and decreasing weight in adolescents with metabolic syndrome
2. To evaluate the tolerability of a non-energy restricted very-low carbohydrate diet in these patients as measured by the SF-10 for Children, the Brief Symptom Inventory (BSI) and a scaled questionnaire regarding side effects.
3. To compare two different maintenance programs in the group who receive the non- energy restricted very-low carbohydrate diet and compare each group to the group

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults ages 13-18 with a BMI>95% for age or over 30 for young adults, with pre-existing metabolic syndrome

Exclusion Criteria:

* Subjects on any chronic medication other than antihistamines, asthma medications, oral contraceptives or diabetes medications, smoke more than 5 cigarettes/day, suffer from alcoholism or drug abuse or have any significant abnormality not associated with metabolic syndrome on screening labs will be excluded from randomization.
* Subjects currently taking Byetta will be excluded from the study, as a side effect of the drug is weight loss.
* Subjects with familial hypercholesteremia may be excluded if the investigator considers the history to be severe. The data collected from subjects with a HBA1C greater than 12.5 will be analyzed in a separate group, although they will still be randomized to one of the three treatment groups. This is due to the fact that past experience has shown that these individuals run a high risk of being non-compliant with medication use, diet, and exercise plans. Results from this group will be reported separately.
* Subjects who are pregnant or those desiring pregnancy will be excluded, as the safety of this intervention in pregnancy has not been established.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
weight loss | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Steven Sondike, MD, Principal Investigator — WVU Department of Pediatrics
Locations (1):
- Wvu Department of Pediatrics, Charleston, West Virginia, United States